CLINICAL TRIAL: NCT03592992
Title: Spinal Hydromorphone Versus Morphine for Post-Cesarean Delivery Analgesia: A Non-Inferiority Trial
Brief Title: Spinal Hydromorphone Versus Morphine for Post-Cesarean Delivery Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4357
Record Dates: First submitted 2018-03-26; First posted 2018-07-19 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Institutional Research Ethics Board Approval was obtained (Western Research Ethics Board 111264). Term pregnant women presenting to the Obstetric Care Unit at Victoria Hospital for an elective cesarean delivery will be approached for recruitment. Consenting participants will be randomly assigned to receive either 75 mcg of hydromorphone or 150 mcg of morphine at the time of their spinal anesthetic. Randomization will be achieved through a simple computerized randomization technique (use of random numbers list for allocation).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Allocation concealment will be achieved through central pharmacy randomization with the use of a master randomization list of computer-generated random numbers prior to initiation of recruitment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Spinal Hydromorphone (Experimental): For the intervention group, 75 mcg of hydromorphone will be added to the spinal anesthetic mixture as a one-time injection prior to cesarean delivery.
  Interventions: Drug: Spinal Hydromorphone
- Spinal Morphine (Active Comparator): For the control group,150 mcg of preservative-free morphine will be added to the spinal anesthetic mixture as a one-time injection prior to cesarean delivery.
  Interventions: Drug: Spinal Morphine

INTERVENTIONS:
Drug: Spinal Hydromorphone — 75 mcg of hydromorphone will be prepared in a non-identifiable syringe by central hospital pharmacy. The resulting solution will then be added to the spinal anesthetic mixture(fentanyl 15 mcg and 0.75% hyperbaric bupivacaine 1.4-1.6 mcg at the discretion of the attending anesthesiologist, adjusted to height and weight)
  Arms: Spinal Hydromorphone
Drug: Spinal Morphine — 150 mcg of morphine will be prepared in a non-identifiable syringe by central hospital pharmacy.The resulting solution will be added to the spinal anesthetic mixture (fentanyl 15 mcg and 0.75% hyperbaric bupivacaine 1.4-1.6 mcg at the discretion of the attending anesthesiologist, adjusted to height and weight)
  Arms: Spinal Morphine

SUMMARY:
Morphine is usually used for pain relief after cesarean delivery. However, sometimes it is not available, the patient might be allergic to morphine or intolerant to its side effects. Hydromorphone, another drug from the same class, might be used alternatively, but we need to prove that it is not inferior to morphine.

DETAILED DESCRIPTION:
Spinal or intrathecal (IT) morphine is the most commonly used opioid for post-cesarean delivery analgesia. Factors that contribute to its widespread use include a favorable pharmacokinetic profile with duration of action up to 24 hours, ease of administration (during spinal block for surgical anesthesia) and low cost. Most providers administer 100 to 200 mcg of IT morphine for cesarean delivery analgesia with excellent analgesic results. Nevertheless, subarachnoid use of morphine is not without adverse events. While dose-dependent respiratory depression is the most worrisome complication, other side effects such as pruritus, nausea, vomiting and urinary retention can be bothersome during early puerperium. Furthermore, shortages of preservative free morphine in the United States has led clinicians to seek a reasonable alternative.

For the last 20 years, spinal hydromorphone has been successfully used for chronic pain associated with neoplasms. Its use for post-cesarean analgesia has been successfully reported. However, data regarding its efficacy in the IT space for post-cesarean analgesia is scarce. In the past, doses of 40 to 100 mcg have been reported to provide adequate postoperative pain relief with minimal side effects. In a recent study, the Effective Dose in 90% of patients has been established for both Hydromorphone and Morphine to be 75 mcg and 150 mcg, respectively.

No prospective studies have been conducted to specifically establish non-inferiority of hydromorphone when compared to morphine for post- cesarean analgesia. In addition, while all opioids share the same side effect profile, the frequency of those events are unknown for IT hydromorphone.

The current proposal is a blinded randomized controlled trial of intrathecal hydromorphone versus morphine in term pregnant women undergoing elective cesarean deliveries under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years; American Society of Anesthesiologist's Physical Status (ASA-PS) < 3; Term pregnancy (> 37 weeks gestational age); Elective cesarean delivery; Spinal Anesthesia;

Exclusion Criteria:

* Documented allergy or severe intolerance to opioids; Intra-operative conversion to a general anesthetic technique; Chronic pain syndrome with baseline pain levels >3 on a visual analogue scale (0-10 cm); History of opioid use during this pregnancy; Allergy or intolerance to NSAIDS or acetaminophen; Morbid obesity- Body Mass Index (BMI) >40.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects that are term pregnant at the time of recruitment.
Enrollment: 126 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Difference in the Average Numeric Rating Score (0-10 , where 0=no pain and 10= maximum pain) during the first 24 hours. | 24 hours after spinal anesthesia.
  This is defined as the between- group difference in the average pain scores on a 0-10 Numeric Rating Scale, as assessed by a nurse, anesthesia consultant or trainee 24 hours after spinal anesthesia.

SECONDARY OUTCOMES:
Difference in NRS pain scores at specific time points in the first 24 hours. | immediately after surgery (in PACU), 6, 12 and 18 hours after spinal anesthesia is given.
  This is defined as the between- group difference in the mean pain scores on a 0-10 Numeric Rating Scale, as assessed by a nurse, anesthesia consultant or trainee immediately after surgery (in the Post-Anesthesia Care Unit) and at 6, 12, 18 and 24 hours after spinal anesthesia.
Time-to-first oral opioid analgesic request | Measured in hours from the time of spinal anesthetic until patient request for prescribed oral opioid analgesia, up to 24 hours from the spinal anesthetic .
  This is defined as the length of time between spinal anesthesia and the first time the subject requested additional opioid analgesia, up to 24 hours from the spinal anesthesia.
Nausea and/or Vomiting that required treatment. | Absolute number of treatments required in the 24-hour time frame.
  Nausea/Vomiting episodes that required pharmacological treatment in the first 24 hours after spinal anesthesia
Pruritus that required treatment. | Absolute number of treatments required in the 24-hour time frame.
  Pruritus episodes that required pharmacological treatment in the first 24 hours after spinal anesthesia
Respiratory Depression | In post-anesthesia care unit (PACU), 6, 12, 18 and 24 hours after spinal anesthesia
  Respiratory Rate measured in breaths/minute)
Apgar Scores | 1 and 5 minutes after birth.
  Neonatal Apgar scores at 1 and 5 minutes in a 1-10 interval scale
Difference in Opioid Consumption in the first 24 hours | 24 hours after spinal anesthesia.
  This is defined as the between-group difference in the total amount of Oral Morphine Equivalents consumed in the first 24 hours after spinal anesthesia is given.
Obstetric Quality of Recovery Score ObsQoR-11 | 24 hours after spinal anesthesia.
  11-item questionnaire applied to subjects 24 hours after spinal anesthesia. Measured in a 0-110 scale

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Sebbag, MD, Principal Investigator — Western University
Locations (1):
- Victoria Hospital- LHSC, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared after the end of this study other than publication of study results in medical journals.

REFERENCES:
- [Background] Palmer CM, Emerson S, Volgoropolous D, Alves D. Dose-response relationship of intrathecal morphine for postcesarean analgesia. Anesthesiology. 1999 Feb;90(2):437-44. doi: 10.1097/00000542-199902000-00018. PMID 9952150
- [Background] Rathmell JP, Pino CA, Taylor R, Patrin T, Viani BA. Intrathecal morphine for postoperative analgesia: a randomized, controlled, dose-ranging study after hip and knee arthroplasty. Anesth Analg. 2003 Nov;97(5):1452-1457. doi: 10.1213/01.ANE.0000083374.44039.9E. PMID 14570664
- [Background] Wong JY, Carvalho B, Riley ET. Intrathecal morphine 100 and 200 mug for post-cesarean delivery analgesia: a trade-off between analgesic efficacy and side effects. Int J Obstet Anesth. 2013 Jan;22(1):36-41. doi: 10.1016/j.ijoa.2012.09.006. Epub 2012 Nov 15. PMID 23159009
- [Background] Milner AR, Bogod DG, Harwood RJ. Intrathecal administration of morphine for elective Caesarean section. A comparison between 0.1 mg and 0.2 mg. Anaesthesia. 1996 Sep;51(9):871-3. doi: 10.1111/j.1365-2044.1996.tb12622.x. PMID 8882255
- [Background] Girgin NK, Gurbet A, Turker G, Aksu H, Gulhan N. Intrathecal morphine in anesthesia for cesarean delivery: dose-response relationship for combinations of low-dose intrathecal morphine and spinal bupivacaine. J Clin Anesth. 2008 May;20(3):180-5. doi: 10.1016/j.jclinane.2007.07.010. PMID 18502360
- [Background] Gerancher JC, Floyd H, Eisenach J. Determination of an effective dose of intrathecal morphine for pain relief after cesarean delivery. Anesth Analg. 1999 Feb;88(2):346-51. doi: 10.1097/00000539-199902000-00023. PMID 9972754
- [Background] Ventola CL. The drug shortage crisis in the United States: causes, impact, and management strategies. P T. 2011 Nov;36(11):740-57. No abstract available. PMID 22346307
- [Background] Deer TR, Smith HS, Burton AW, Pope JE, Doleys DM, Levy RM, Staats PS, Wallace MS, Webster LR, Rauck RL, Cousins M; Center For Pain Relief, Inc. Comprehensive consensus based guidelines on intrathecal drug delivery systems in the treatment of pain caused by cancer pain. Pain Physician. 2011 May-Jun;14(3):E283-312. PMID 21587338
- [Background] Dougherty TB, Baysinger CL, Henenberger JC, Gooding DJ. Epidural hydromorphone with and without epinephrine for post-operative analgesia after cesarean delivery. Anesth Analg. 1989 Mar;68(3):318-22. PMID 2465709
- [Background] Parker RK, Sawaki Y, White PF. Epidural patient-controlled analgesia: influence of bupivacaine and hydromorphone basal infusion on pain control after cesarean delivery. Anesth Analg. 1992 Nov;75(5):740-6. doi: 10.1213/00000539-199211000-00015. PMID 1384397
- [Background] Beatty NC, Arendt KW, Niesen AD, Wittwer ED, Jacob AK. Analgesia after Cesarean delivery: a retrospective comparison of intrathecal hydromorphone and morphine. J Clin Anesth. 2013 Aug;25(5):379-383. doi: 10.1016/j.jclinane.2013.01.014. Epub 2013 Aug 17. PMID 23965210
- [Background] Rauch E. Intrathecal hydromorphone for postoperative analgesia after cesarean delivery: a retrospective study. AANA J. 2012 Aug;80(4 Suppl):S25-32. PMID 23248827
- [Background] Sviggum HP, Arendt KW, Jacob AK, Niesen AD, Johnson RL, Schroeder DR, Tien M, Mantilla CB. Intrathecal Hydromorphone and Morphine for Postcesarean Delivery Analgesia: Determination of the ED90 Using a Sequential Allocation Biased-Coin Method. Anesth Analg. 2016 Sep;123(3):690-7. doi: 10.1213/ANE.0000000000001229. PMID 26974022
- [Background] Rauch E. Intrathecal hydromorphone for cesarean delivery: in search of improved postoperative pain management: a case report. AANA J. 2011 Oct;79(5):427-32. PMID 23256273
- [Background] Ciechanowicz S, Setty T, Robson E, Sathasivam C, Chazapis M, Dick J, Carvalho B, Sultan P. Development and evaluation of an obstetric quality-of-recovery score (ObsQoR-11) after elective Caesarean delivery. Br J Anaesth. 2019 Jan;122(1):69-78. doi: 10.1016/j.bja.2018.06.011. Epub 2018 Jul 31. PMID 30579408
- [Derived] Cheng S, Bartolacci J, Armstrong K, Dobrowlanski A, Jones PM, Singh SI, Sebbag I. Intrathecal Hydromorphone Versus Intrathecal Morphine for Postcesarean Delivery Analgesia: A Randomized Noninferiority Trial. Anesth Analg. 2026 Jan 1;142(1):19-27. doi: 10.1213/ANE.0000000000007580. Epub 2025 Jun 10. PMID 40493496